CLINICAL TRIAL: NCT03111355
Title: Genetic Variants in Selenoprotein Genes and Gender Influence Biomarkers of Se Status in Response to Brazil Nut Supplementation in Healthy Brazilians
Brief Title: Effects of Genetic Variations in the Response to Brazil Nut Supplementation
Acronym: SUBRANUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Newcastle University (Other); University of Aberdeen (Other); Aix Marseille Université (Other)
Responsible Party: Principal Investigator, Janaina Donadio, Principal Investigator, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: USPBR
Record Dates: First submitted 2017-03-27; First posted 2017-04-12 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Dietary Supplements
Keywords: nuts; micronutrients; nutrigenomics; nutrigenetics
MeSH Terms: interventions — 2S albumin, brazil nut

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brazil Nut supplementation (Experimental): Consumption of one Brazil nut a day for 2 months followed by 2 months without intervention
  Interventions: Dietary Supplement: Brazil nut

INTERVENTIONS:
Dietary Supplement: Brazil nut — one nut a day for 2 months, no intervention for 2 months

SUMMARY:
This study investigates the effect of genetic variations after supplementation with Brazil nuts in healthy Brazilians. Briefly, all the participants will consume one nut a day for 2 months and will stop the intake for more 2 months. Five blood sampling collection will be performed in one month interval, starting at baseline and ending at 2 months without intervention.

DETAILED DESCRIPTION:
Brazil nuts are the richest source of selenium in nature, a micronutrient that has essential functions in human physiology.

Selenium status can be measured by the quantification of biomarkers in the blood. Previous studies have shown that genetic polymorphisms can affect Se status and modulate risk for chronic diseases. In this study, five biomarkers will be quantified in the blood, before and after supplementation with Brazil nuts. The genetic variants will be used to stratify the biomarkers and multivariate linear regressions will be used to explore the influence of the polymorphisms on concentrations of the biomarkers .

ELIGIBILITY:
Inclusion Criteria:

* age between 20 and 60 years; not taking vitamin and minerals supplements, not taking antiinflammatory, not having chronic diseases

Exclusion Criteria:

* athletes, excessive alcohol consumption, being obese, having cancer, cardiovascular disease, diabetes and hypo or hyperthyroidism

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2014-08-15 (Actual); Study Completion 2016-04-19 (Actual)

PRIMARY OUTCOMES:
change in Plasma Se concentrations | 4 weeks
  measured by ICP-MS (ug/L)
change in Plasma Glutathione Peroxidase 3 activity | 4 weeks
  measured by kinetic assay in a spectrometer (U/L)
change in Plasma Selenoprotein P concentrations | 4 weeks
  measured by ELISA (mg/dL)
change in Erythrocyte Se concentrations | 4 weeks
  measured by ICP-MS (ug/L)
change in Erythrocyte Glutathione Peroxidase 1 activity | 4 weeks
  measured by kinetic assay in an automatic spectrometer (U/gHb)

SECONDARY OUTCOMES:
change in total cholesterol concentration in serum | 4 weeks
  measured in an automatic spectrometer (mg/dL)
change in tryglicerides concentration in serum | 4 weeks
  measured in an automatic spectrometer (mg/dL)
change in HDL concentration in serum | 4 weeks
  measured in an automatic spectrometer (mg/dL)
change in LDL concentration in serum | 4 weeks
  measured in an automatic spectrometer (mg/dL)
change in protein-c reactive concentration in serum | 4 weeks
  measured in an automatic spectrometer (mg/dL)
change in Plasma MDA concentrations (malondialdehyde) | 4 weeks
  measured in an automatic spectrometer (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia MF Cozzolino, PhD, Principal Investigator — University of Sao Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Donadio JL, Guerra-Shinohara EM, Rogero MM, Cozzolino SM. Influence of Gender and SNPs in GPX1 Gene on Biomarkers of Selenium Status in Healthy Brazilians. Nutrients. 2016 May 5;8(5):81. doi: 10.3390/nu8050081. PMID 27164132
- [Result] Donadio JLS, Rogero MM, Guerra-Shinohara EM, Desmarchelier C, Borel P, Cozzolino SMF. SEPP1 polymorphisms modulate serum glucose and lipid response to Brazil nut supplementation. Eur J Nutr. 2018 Aug;57(5):1873-1882. doi: 10.1007/s00394-017-1470-7. Epub 2017 May 13. PMID 28501922
- [Result] Donadio JLS, Rogero MM, Cockell S, Hesketh J, Cozzolino SMF. Influence of Genetic Variations in Selenoprotein Genes on the Pattern of Gene Expression after Supplementation with Brazil Nuts. Nutrients. 2017 Jul 11;9(7):739. doi: 10.3390/nu9070739. PMID 28696394
- [Result] Donadio JLS, Rogero MM, Guerra-Shinohara EM, Barbosa F Jr, Desmarchelier C, Borel P, Sneddon AA, Hesketh JE, Cozzolino SMF. Genetic variants in selenoprotein genes modulate biomarkers of selenium status in response to Brazil nut supplementation (the SU.BRA.NUT study). Clin Nutr. 2019 Apr;38(2):539-548. doi: 10.1016/j.clnu.2018.03.011. Epub 2018 Mar 23. PMID 29609868